CLINICAL TRIAL: NCT05389813
Title: Comparison Between Oxycodone and Pregabalin as Preemptive Analgesia for Postoperative Pain Control, Placebo-controlled RCT, 2021
Brief Title: Comparison Between Oxycodone and Pregabalin as Preemptive Analgesia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: An-Najah National University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Preemptive Analgesia
Record Dates: First submitted 2022-02-15; First posted 2022-05-25 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Anesthesia
MeSH Terms: interventions — Oxycodone; Tablets; Pregabalin; Geritol; Minerals

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Oxycodone (Active Comparator): 20 mg oxycodone hydrochloride and 10 mg naloxone hydrochloride given as 1 tablet only once, 30 minutes preoperatively.
  Interventions: Drug: Oxycodone 20 Mg Oral Tablet
- Pregabalin (Active Comparator): 150 mg Pregabalin given as 1 tablet only once, 30 minutes preoperatively.
  Interventions: Drug: Pregabalin 150mg
- Multivitamin (Placebo Comparator): Abecedin Multivitamins&Minerals given as 1 tablet only once, 30 minutes preoperatively.
  Interventions: Drug: Multivitamin with Minerals

INTERVENTIONS:
Drug: Oxycodone 20 Mg Oral Tablet — Oxycodone is a semi-synthetic, morphine-like opioid alkaloid with analgesic activity. Oxycodone exerts its analgesic activity by binding to the mu-receptors in the central nervous system (CNS), thereby mimicking the effects of endogenous opioids. Binding of the opiate receptor stimulates the exchange of GTP for GDP on the G-protein complex and inhibits adenylate cyclase, thereby preventing cAMP production. Subsequently, the release of nociceptive neurotransmitters, such as substance P, gamma-aminobutyric acid (GABA), dopamine, acetylcholine, and noradrenaline, is inhibited. Oxycodone also inhibits the release of vasopressin, somatostatin, insulin, and glucagon. In addition, oxycodone closes N-type voltage-gated calcium channels and opens G-protein-coupled inwardly rectifying potassium channels resulting in hyperpolarization and reduction of neuronal excitability.
  Other Names: Targin
  Arms: Oxycodone
Drug: Pregabalin 150mg — Pregabalin is a gabapentinoid and acts by inhibiting certain calcium channels. Specifically it is a ligand of the auxiliary α2δ subunit site of certain voltage-dependent calcium channels (VDCCs), and thereby acts as an inhibitor of α2δ subunit-containing VDCCs. There are two drug-binding α2δ subunits, α2δ-1 and α2δ-2, and pregabalin shows similar affinity for (and hence lack of selectivity between) these two sites. Pregabalin is selective in its binding to the α2δ VDCC subunit. Despite the fact that pregabalin is a GABA analogue. r synthesizing GABA, and hence may have some indirect GABAergic effects by increasing GABA levels in the brain. In accordance, inhibition of α2δ-1-containing VDCCs by pregabalin appears to be responsible for its anticonvulsant, analgesic, and anxiolytic effects.
  Other Names: Lyrica
  Arms: Pregabalin
Drug: Multivitamin with Minerals — Vit A 3000 IU, Vit B1 2.5mg, Vit B2 2.0mg, Vit B12 10mcg, Vit C 150mg, Vit D3 400 IU, Vit E10 IU, Biotin 25mcg, Nicotimamide 30mg, Calcium Pantothenate 3mg, Folic acid 800mcg, Iron Fumarate 18mg, Calcium 125mg, Magnesium Oxide 10mg, Iodine Potassium 150mcg, Manganese sulfate 0.5mg, Phosphorus 23.8mg, Copper sulfate 1.0mg, Molybdinium Sodium 0.10mg, Zinc Sulfate 5.0mg.
  Other Names: Abecedin
  Arms: Multivitamin

SUMMARY:
The research will be conducted between March 2021 and June 2023. All patients scheduled electively for one of four surgeries (Laparoscopic Cholecystectomy, Submucosal resection, Breast lumpectomy, and median laparotomy) at that period of time at An-Najah National University hospital will be included in the research sample, unless not meeting with the criteria put.

Primary objectives are:

To evaluate the effectiveness of preemptive analgesia on postoperative pain relief and shorter hospital stay for adults undergoing surgical procedures, according to the type of surgery and the type of drug.

To compare the effect of a single oral preemptive dose of Pregabalin versus Oxycodone on postoperative pain relief, in terms of pain intensity as assessed by pain numeric rating scale (NRS)

DETAILED DESCRIPTION:
* After signing the informed consent, each participant will undergo standard care for any surgical patient (general examination, vital signs recording, history taking, and cannula insertion). Then, a nurse will teach him\her how to use the NRS for pain scores.
* Patients will be randomly allocated by computer-generated list to Group A (oxycodone 20 mg orally), Group B (pregabalin 150 mg orally), or Group C (multivitamins pill orally).
* The medication will be given 30 minutes before operation by an anesthesiology resident who is not aware of the study design in a closed envelope with a code similar to the file code of the participant and he will make sure that the participant ingests the pill with a sip of water and get rid of the envelope immediately.
* The participant then will be transferred to the preparation room before surgery, baseline scores will be recorded for the following parameter: pain scale (NRS) during rest and movement, Modified Ramsay Sedation Score (MRSS), and vital signs.
* Patient then will be transferred to the operation room, and induction of anaesthesia will begin.

The anaesthetic protocol will be standardized.

* The anaesthetists will record the duration of surgery as the time between induction of anaesthesia and arrival to Post-Anesthetic Care Unit (PACU). Arrival to PACU will be recorded as 0 times.
* The participant will be sent to the ward after collecting 8 points or greater or return to baseline on Post-Anesthesia Recovery Score (PARS). Time in PACU will be reported.
* A postoperative patient evaluation will be performed by an anaesthetist who will be unaware of the study design.
* Postoperative pain treatment will be with patient-controlled IV morphine 2.5 mg bolus (rescue analgesia). Nausea will be treated with ondansetron.
* Morphine consumption, pain intensity at rest and during mobilization, nausea and vomiting, sedation, dizziness, and consumption of ondansetron will be recorded at 0, 1, 4, and 8 h after operation.
* On discharge, time and date of discharge and satisfaction of analgesia score will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18-year-old.
2. Patients undergoing elective surgeries under general anesthesia.
3. American Society of Anesthesiology grade 1 or 2.
4. BMI 18-35 Kg/m2
5. Reliable participant (he/she can give history by him/herself)

Exclusion Criteria:

1. Current Pregnancy or breastfeeding.
2. Chronic use of analgesia (use of any analgesic drug for most days in the last three months).
3. Current use of analgesia (within last 24 hours).
4. Allergy to any medication used in the study.
5. Smoking or Nargila use within last 24 hour before surgery and until discharge.
6. History of psychiatric medication or disease.
7. Discharge from hospital within 6 hours after surgery.
8. Participants transferred from the ward to ICU or other wards.
9. Known case of liver or kidney impairment.
10. History of alcohol use or illicit drug.
11. Any complication during surgery leads to changes in protocol of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative pain | 30 minutes preoperative
  The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"), has become the most widely used instrument for pain screening. This will have 2 contents:
  * NRS at rest.
  * NRS at movement.
Postoperative pain | at 0 hour postoperative
  The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"), has become the most widely used instrument for pain screening.
Postoperative pain | at 1 hour postoperative
  The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"), has become the most widely used instrument for pain screening.
Postoperative pain | at 4 hour postoperative
  The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"), has become the most widely used instrument for pain screening.
Postoperative pain | at 8 hour postoperative
  The pain numeric rating scale (NRS), on which patients rate their current pain intensity from 0 ("no pain") to 10 ("worst possible pain"), has become the most widely used instrument for pain screening.

SECONDARY OUTCOMES:
Sedation | 30 minutes preoperative, at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  Using the eight-point Modified Ramsay Sedation Score:
  1. Awake and alert, minimal or no cognitive impairment.
  2. Awake but tranquil, purposeful responses to verbal commands at a conversational level.
  3. Appears asleep, purposeful response to verbal commands at a conversational level.
  4. Appears asleep, purposeful responses to commands but at a louder than conversational level, requiring light glabellar tap, or both.
  5. Asleep, sluggish purposeful responses only to loud verbal commands, strong glabellar tap, or both.
  6. Asleep, sluggish purposeful responses only to painful stimuli.
  7. Asleep, reflex withdrawal to painful stimuli only
  8. Unresponsive to external stimuli, including pain
Heart rate | 30 minutes preoperative, at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  it will be measured by pulse oximeter and expressed as beats per minute.
Respiratory rate | 30 minutes preoperative, at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  it will be measured by counting the number of breaths for one minute by counting how many times the chest rises and expressed as breaths per minute.
Temperature | 30 minutes preoperative, at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  it will be measured by thermometer and expressed in degrees Celsius ( °C ).
Blood pressure | 30 minutes preoperative, at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  Systolic and diastolic blood pressure will be measured by sphygmomanometer and expressed in millimeters of mercury (mmHg).
O2 saturation | 30 minutes preoperative, at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  it will be measured by pulse oximeter and expressed as percent (%).
Drug side effects | at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  Measuring the incidence of undesirable effect of a drug (constipation, respiratory depression, diarrhea, headache, dyspepsia, itching, urinary retention, and pruritus) using a questionnaire with Yes or No answer.
Postoperative nausea and vomiting | At 6 hour postoperative
  Postoperative nausea and vomiting intensity scale Q1 Have you vomited or had dry-retching?
  1. No(0-Score)
  2. Once or twice(2-Score)
  3. Three or more times(50-Score) Q2 Have you experienced a feeling of nausea (an unsettled feeling in the stomach and slight urge to vomit)? If yes. has your feeling of nausea interfered with activities of daily living? such as being able to get out of bed, being able to move about freely in bed, being able to walk normally or eating and drinking?
  a) No(0-Score) b) Sometimes(1-Score) c) Often or most of the time(2-Score) d) All of the time(25-Score)
  Q3 Has your nausea been mostly:
  1. varying?(1-Score)
  2. constant?(2-Score) Q4 What was the duration of your feeling of nausea(in hours)? Where a score ≥50 defined clinically important PONV: PONV Intensity Scale=severity of nausea (1=mild, 2=moderate, 3=severe) × pattern of nausea (1=varying, 2=constant) × duration of nausea (in hours)
Rescue analgesia | at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  Time to first use of rescue analgesia (which is 3 my IV Morphine) and Total analgesic consumption (mg/kg)
Antiemetics | at 0 hour postoperative, at 1 hour postoperative 4, at 8 hour postoperative.
  Time to first use of antiemetics (which is 4 mg IV Ondansetrone) and Total analgesic consumption (mg/kg)

CONTACTS AND LOCATIONS:
Overall Officials: Zaher Nazzal, Study Director — An-Najah National University
Locations (1):
- An-Najah National University Hospital, Nablus, Wes-Bank, Palestinian Territories